CLINICAL TRIAL: NCT07181174
Title: Renal Resistive Index as a Predictor of Acute Kidney Injury in Patient With Hemorrhagic Stroke
Brief Title: Early Prediction and Diagnosis of Acute Kidney Injury
Status: Enrolling by invitation | Type: Observational
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Peter Essa, Resident of neuropsychiatry department, Aswan University
Other Study IDs: 1016/11/24
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Early Diagnosis of Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Ultrasonographic examination and doppler ultrasonography will be performed using a convex transducer. — -Renal Resistive Index Measurement Method: Ultrasonographic examination and doppler ultrasonography will be performed using a convex transducer. First, the kidney is localised in the flanks with conventional B-mode ultrasonography, after which, color doppler images are acquired. The interlobar arteries were visualised, with the wavelength obtained by creating a 90-degree right-angle with the interlobar artery using a power doppler. After the manual determination of the peak systolic and end-diastolic velocities * RRI will be calculated by the device using the formula: RRI = (peak systolic velocity - end-diastolic velocity) / (peak systolic velocity). RRI will be measured three times for each kidney and averaged

SUMMARY:
The goal of this clinical trial is to estimate the accuracy of renal resistive index in early diagnosis and prediction of acute kidney injury in patients with hemorrhagic stroke. the main questions it aims to answer are :

* Early detection of acute kidney injury in patient with hemorrhagic stroke .
* Decrease morbidity and mortality rate in patients with hemorrhagic stroke .

ELIGIBILITY:
Inclusion Criteria:

All patients with hemorrhagic stroke presented to Aswan university hospital that will be fulfilled the following characters:

* Age >18 years.
* Both sex.
* Cases of spontaneous onset

Exclusion Criteria:

* Age < 18
* Patients with traumatic hemorrhagic stroke.
* Patients with brain tumors.
* Patients with congenital anomalies of cerebral vessels e.g. AVM (arteriovenous malformation) and cerebral aneurysm.
* Patients with history of any renal diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with hemorrhagic stroke
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Early detection of acute kidney injury in patient with hemorrhagic stroke | within 2 days and 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan university hospitals- Neurology Department, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No